CLINICAL TRIAL: NCT05728905
Title: Effects on Pain and Function When Implementing an Orthopedic Manual Therapy Intervention Compared to an Exercise Program Intervention in Patients With Painful Disc Displacement With Reduction
Brief Title: Effects on Pain and Function of Orthopedic Manual Therapy in Patients With Painful Disc Displacement With Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisioterapia Manual Ortopedica (Network)
Responsible Party: Principal Investigator, ARMANDO CAMPOS, Director, Fisioterapia Manual Ortopedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMO Fisioterapia
Record Dates: First submitted 2022-07-25; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Temporomandibular Disorder; Manual Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Exercise Therapy; Exercise; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A randomized single blind clinical trial
Who Masked: Outcomes Assessor
Masking Description: The assessing physiotherapist did not know to which group the patient belongs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic exercise (Experimental): The patients assigned to this group performed a self-treatment program that included three coordination exercises, two post-isometric relaxation (contraction-relaxation) and one self-traction. All exercises were performed in front of a mirror. It was performed every 3 hours, 5 times a day, for 4 weeks. The patient was instructed and supervised by a physiotherapist until they were executed correctly. All participants were provided with a video where the procedure and dosage of each exercise was described in detail.
  Interventions: Other: Therapeutic exercise
- Therapeutic exercise + orthopedic manual therapy (Experimental): The patients assigned to this group performed the exercise program and also received a manual therapy treatment applied by a physiotherapist. Two sessions were held per week for 4 weeks (8 sessions). Treatment consisted of traction, mobilization, and friction massage of the muscles of mastication.
  Interventions: Other: Therapeutic exercise; Other: Orthopedic manual therapy
- Control (No Intervention): The patients assigned to this group did not receive any type of intervention during the 4 weeks. They were asked not to change their habits or receive any other type of treatment.

INTERVENTIONS:
Other: Therapeutic exercise — Intervention with therapeutic exercise: coordination, relaxation and disc recapture exercises.
  Other Names: Exercise
  Arms: Therapeutic exercise; Therapeutic exercise + orthopedic manual therapy
Other: Orthopedic manual therapy — Intervention with orthopedic manual therapy: traction, ventral sliding and massage.
  Other Names: Physiotherapy
  Arms: Therapeutic exercise + orthopedic manual therapy

SUMMARY:
The objective of this study was to compare the short- and medium-term effects in pain and temporomandibular joint (TMJ) and function of implementing a manual therapy (MT) intervention treatment combined with a therapeutic exercise (TE) program, versus an isolated TE program and a non-intervention in patients with disc displacement with reduction (DDCR) with pain.

DETAILED DESCRIPTION:
Study Design: The study adopted a single-blind, randomized, controlled clinical trial approach. Adults with disc displacement with reduction clinical diagnosis, pain and loss of function were eligible for inclusion.

Intervention: Patients in the study were randomized into three groups, 25 subjects to the manual therapy and therapeutic exercise group, 25 to the therapeutic exercise group and 25 to the no intervention group. Subjects were excluded if there was presence of surgical history, dentistry treatment and use of medication. The dependent variables were the presence of clicking, TMJ function, cervical disability, pain, and range of motion of the TMJ. Subjects in every group were assessed after four weeks of intervention and after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Disc displacement with reduction diagnosis according to the Research Diagnostic Criteria for Temporomandibular Disorders; in the last 30 days, any TMJ noise present during the exam or clicking detected with palpation during at least one of three repetitions of jaw opening, closing, protrusion, or laterotrusion movements.
* equal or greater than 30 mm on the VAS scale
* Age is greater than or equal to18 years.

Exclusion Criteria:

* Participants were excluded if they had received interventions of TMJ surgery or TMJ steroid injections in the previous month, a rheumatoid diagnosis, neurological or psychiatric diseases, or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Effects on pain when implementing an orthopedic manual therapy intervention compared to an exercise program intervention in patients with painful disc displacement with reduction | 3 months
  Pain prevalence within patients with disc displacement, evaluated using Visual Analogue Scale (VAS).
Effects on function when implementing an orthopedic manual therapy intervention compared to an exercise program intervention in patients with painful disc displacement with reduction | 3 months
  Prevalence of jaw disfunction in patients with disc displacement, assessed using Jaw Functional Limitation Scale-20.

CONTACTS AND LOCATIONS:
Overall Officials: ARMANDO CAMPOS, Principal Investigator — FMO
Locations (1):
- Clinic, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au AR, Klineberg IJ. Isokinetic exercise management of temporomandibular joint clicking in young adults. J Prosthet Dent. 1993 Jul;70(1):33-9. doi: 10.1016/0022-3913(93)90034-l. PMID 8366455
- [Background] Yoda T, Sakamoto I, Imai H, Honma Y, Shinjo Y, Takano A, Tsukahara H, Morita S, Miyamura J, Yoda Y, Sasaki Y, Tomizuka K, Takato T. A randomized controlled trial of therapeutic exercise for clicking due to disk anterior displacement with reduction in the temporomandibular joint. Cranio. 2003 Jan;21(1):10-6. doi: 10.1080/08869634.2003.11746226. PMID 12555926
- [Background] Wanman A, Marklund S. Treatment outcome of supervised exercise, home exercise and bite splint therapy, respectively, in patients with symptomatic disc displacement with reduction: A randomised clinical trial. J Oral Rehabil. 2020 Feb;47(2):143-149. doi: 10.1111/joor.12888. Epub 2019 Sep 30. PMID 31520538
- [Background] Armijo-Olivo S, Pitance L, Singh V, Neto F, Thie N, Michelotti A. Effectiveness of Manual Therapy and Therapeutic Exercise for Temporomandibular Disorders: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jan;96(1):9-25. doi: 10.2522/ptj.20140548. Epub 2015 Aug 20. PMID 26294683
- [Background] Craane B, Dijkstra PU, Stappaerts K, De Laat A. Randomized controlled trial on physical therapy for TMJ closed lock. J Dent Res. 2012 Apr;91(4):364-9. doi: 10.1177/0022034512438275. Epub 2012 Feb 8. PMID 22318373
- [Background] Campos Lopez A, De-Miguel EE, Malo-Urries M, Acedo TC. Mouth opening, jaw disability, neck disability, pressure pain thresholds, and myofascial trigger points in patients with disc displacement with reduction: A descriptive and comparative study. Cranio. 2024 May;42(3):309-315. doi: 10.1080/08869634.2021.1956214. Epub 2021 Aug 12. PMID 34382921
- [Background] Medlicott MS, Harris SR. A systematic review of the effectiveness of exercise, manual therapy, electrotherapy, relaxation training, and biofeedback in the management of temporomandibular disorder. Phys Ther. 2006 Jul;86(7):955-73. PMID 16813476
- [Result] Tuncer AB, Ergun N, Tuncer AH, Karahan S. Effectiveness of manual therapy and home physical therapy in patients with temporomandibular disorders: A randomized controlled trial. J Bodyw Mov Ther. 2013 Jul;17(3):302-8. doi: 10.1016/j.jbmt.2012.10.006. Epub 2012 Nov 16. PMID 23768273